CLINICAL TRIAL: NCT04065750
Title: Exposure to Antibiotics and Incidence of Bacteraemia Caused by Resistant Bacteria
Acronym: BactHub
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Versailles Saint-Quentin-en-Yvelines University (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190295
Record Dates: First submitted 2019-08-19; First posted 2019-08-22 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Bacteremia
Keywords: bacteremia; resistant bacteria; antibiotic
MeSH Terms: conditions — Bacteremia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of the study is to identify the risk factors of community-acquired bacteremia to resistant bacteria.

As the secondary objectives, the study aims

* to describe the episodes of epidemiology of bacteremia (community-acquired and nosocomial) with inpatient patients in APHP.
* to research a potential correlation between the incidence of community-acquired bacteremia of studied germs and the evolution of antibiotics consumption in general population in Île de France region.
* to distinguish three categories of community-acquired bacteremia: real community-acquired infections, infections beginning in community (patients discharged a community care center within 3 months), the nosocomial infections (patients discharged a health center within 7 jours). Describe the epidemiology of resistance and the differential impact of individual exposure to antibiotics in these three categories.
* to identify, according to pathogens, a temporal threshold from which a prior stay in a health center or HAD would impact on the occurrence of a community-acquired bacteremia with a resistant bacterium.
* to describe prospectively for follow-up of 1 year for hospitalized patients for a community-acquired or nosocomial bacteremia: mortality at one month and 3 months, re-hospitalization for an infectious episode and isolated bacteria during this later episode.

DETAILED DESCRIPTION:
The investigators will study in particularly individual exposure to antibiotics: exposure in 3 months ou in 12 months, cumulative exposure, hospital- and community-acquired exposure, etc.

ELIGIBILITY:
Inclusion Criteria:

For bacteraemia cohort:

All inpatient patients in a hospital of APHP between January 2010 and december 2018 with at least one haemoculture positive.

* presence of at least a bacteremia as primary diagnosis, related diagnosis and associated diagnosis: A40 (streptococcus), A41 (staphylococcus, BGN, anaerobes, others), A32.7 (Listeria), A39.4 (meningocoele), A42.7 (Actinomyces), A02.1 (Salmonella), A54.8 (gonocoque), A48.0 (Clostridium).
* and/or in biological data presence of at least a haemoculture positive to Staphylococcus aureus, Klebsiella pneumoniae, Escherichia coli, Acinetobacter Baumannii, Enterococcus faecium, Enterococcus faecalis, Enterobacter cloacae, Pseudomonas aeruginosa, Streptococcus sp., Salmonella sp., Clostridium difficile.

For control cohort:

Patients cared in a hospital of APHP between 2010 and 2018 without infection. - Patients without infection of CIM-10 bacteraemia as primary diagnosis, related diagnosis and associated diagnosis, without haemoculture positive in microbiology.

Exclusion Criteria:

- Patients aged < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bacteremia cohort: all inpatient patients in a hospital of APHP between January 2010 and december 2018 with at least one haemoculture positive.
  Control cohort: patients cared in a hospital of APHP between 2010 and 2018 without infection.
Sampling Method: Non-Probability Sample
Enrollment: 45000 (Estimated)
Dates: Start 2023-11-13 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of bacteraemia | through study completion, an average of 3 months

SECONDARY OUTCOMES:
Mortality | at 30 day and 90 day
  Events of death will be recorded, the mortality rate will be calculated for 30 day and 90 day.
Rehospitalization | 12 months
  The rate of 12 months unplanned rehospitalization for infection by the same biological pathogenes was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Watier, PhD, Study Director — INSERM / Institut Pasteur; Didier Guillemont, MD, PhD, Principal Investigator — APHP, Université de Versailles Saint-Quentin-en-Yvelines

IPD SHARING:
Plan to Share IPD: No